CLINICAL TRIAL: NCT06161974
Title: Phase 2 Study of Olutasidenib with Temozolomide As Maintenance Therapy in Pediatric and Young Adult Patients Newly Diagnosed with High-Grade Glioma (HGG), Including Diffuse Intrinsic Pontine Glioma (DIPG), Which Harbor IDH1 Mutations
Brief Title: Study of Olutasidenib and Temozolomide in HGG
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TarGeT-D
Record Dates: First submitted 2023-11-22; First posted 2023-12-08 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: High Grade Glioma; Astrocytoma; Astrocytoma, Grade III; Astrocytoma, Grade IV; Diffuse Intrinsic Pontine Glioma; WHO Grade III Glioma; WHO Grade IV Glioma; Metastatic Brain Tumor; Diffuse Midline Glioma, H3 K27M-Mutant; Thalamus Tumor; Spinal Tumor; IDH1 Mutation; IDH1 R132; IDH1 R132C; IDH1 R132H; IDH1 R132S; IDH1 R132G; IDH1 R132L; Oligodendroglioma
MeSH Terms: conditions — Glioma; Astrocytoma; Glioblastoma; Diffuse Intrinsic Pontine Glioma; Brain Neoplasms; Spinal Cord Neoplasms; Oligodendroglioma | interventions — olutasidenib; Temozolomide

STUDY DESIGN:
Intervention Model Description: Olutasidenib +TMZ
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Stratum A (Experimental): Patients with localized, intracranial, non-pontine, and non-thalamic IDH 1 mutant Astrocytoma, CNS WHO Grade 3.
  Interventions: Drug: Olutasidenib + TMZ
- Stratum B (Experimental): Patients with localized, intracranial, non-pontine, and non-thalamic IDH 1 mutant Astrocytoma, CNS WHO Grade 4.
  Interventions: Drug: Olutasidenib + TMZ
- Stratum C (Experimental): Patients with IDH-1 mutant DIPG, primary thalamic and spinal cord IDH-1 mutant HGG.
  Interventions: Drug: Olutasidenib + TMZ

INTERVENTIONS:
Drug: Olutasidenib + TMZ — Olutasidenib 150 mg PO BID + Temozolomide 200 mg/m2 PO QD

SUMMARY:
The goal of this study is to determine the efficacy of the study drug olutasidenib to treat newly diagnosed pediatric and young adult patients with a high-grade glioma (HGG) harboring an IDH1 mutation.

The main question the study aims to answer is whether the combination of olutasidenib and temozolomide (TMZ) can prolong the life of patients diagnosed with an IDH-mutant HGG.

DETAILED DESCRIPTION:
This is a multicenter, international, phase II study of post-radiotherapy (RT) administration of olutasidenib to treat pediatric and young adult patients newly diagnosed with an IDH1-mutant HGG. The trial will include a feasibility cohort to identify the dose of olutasidenib that is feasible when given in combination with temozolomide as maintenance therapy after completion of focal radiotherapy in this patient population.

Efficacy will be defined by progression-free survival (PFS) distribution of these patients after completion of radiotherapy treated with maintenance olutasidenib and TMZ for 13 cycles followed by 13 cycles of single agent olutasidenib compared to molecularly-stratified and matched historical controls.

Objective radiographic response rates, agent-specific toxicities as well as the pharmacokinetic and pharmacodynamic properties of olutasidenib will also be assessed.

ELIGIBILITY:
Criteria TarGeT-D study strata definitions

* Stratum A: Patients with localized, intracranial, non-pontine, and non-thalamic IDH 1 mutant Astrocytoma, CNS WHO Grade 3.
* Stratum B: Patients with localized, intracranial, non-pontine, and non-thalamic IDH 1 mutant Astrocytoma, CNS WHO Grade 4.
* Stratum C: Patients with IDH-1 mutant DIPG, primary thalamic and spinal cord IDH-1 mutant HGG.

Inclusion Criteria:

1. Inclusion criteria already met to enroll on TarGeT-SCR (central molecular and histopathologic screening) based on:

   1.1) Age: patients must be ≥12 years and ≤39 years of age at the time of enrollment on TarGeT-SCR

   1.2) Diagnosis:
   * Patients with a newly-diagnosed IDH1-mutant HGG including DIPG are eligible. All patients must have tumor tissue from diagnostic biopsy or resection, without exceptions. The diagnosis of HGG, including DIPG, must have been confirmed through TarGeT-SCR.
   * For the diagnosis of DIPG, patients must have a tumor with pontine epicenter and diffuse involvement of at least 2/3 of the pons, and histopathology consistent with diffuse WHO Grade 2-4 glioma.
   * All other HGG must be WHO Grade 3 or 4.

   1.3) Disease status: There are no disease status requirements for enrollment
   * Measurable disease is not required. Patients without measurable disease are eligible.
   * Primary spinal tumor: Patients with a primary spinal HGG are eligible.
   * Patient must not have metastatic disease.
2. Inclusion criteria for assignment to TarGeT-D, for all strata:

2.1 Presence of at Least One Relevant Actionable Somatic Mutation in IDH1 Gene, Detailed Here:

* R132H, R132C, R132S, R132G or R132L.
* Patients whose tumors harbor other alterations in addition to IDH1 mutation will potentially be eligible following consensus recommendation by the international multidisciplinary molecular screening committee.
* Patients with IDH2 mutations are not eligible.
* Patients with oligodendroglioma, IDH-mutant and 1p/19q-codeleted are not eligible.

2.2 Performance Level: Karnofsky ≥ 50% for patients > 16 years of age and Lansky ≥ 50 for patients ≤ 16 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

2.3 Prior Therapy

2.3.1 Surgery, radiation, and/or dexamethasone are permissible. Temozolomide administered concurrently with radiotherapy is permissible. No other prior anticancer therapy for HGG will be allowed.

2.3.2 Radiation therapy requirements: RT, delivered via photon or proton beam, must have been administered at a standard dose including 54 Gy in 30 fractions for DIPG, 59.4 Gy in 33 fractions or 54-60 Gy in 30 fractions for other HGG or 45-50.4 Gy for primary spinal disease. Any variances in the radiotherapy dose within 10% of the standard doses outlined above will be discussed with the Study Chair to confirm eligibility prior to study enrollment.

2.3.3 Timing between diagnosis and start of RT: Patients must have started RT within 31 calendar days of initial diagnosis defined as the date of diagnostic biopsy or resection; if a patient underwent two upfront surgeries (e.g., biopsy then resection or debulking), this is the date of the second surgery.

2.3.4 Timing post-RT

* Patients in pre-maintenance phase must enroll and start treatment no later than 21 calendar days post-completion of RT.
* Patients not in pre-maintenance phase must enroll and start treatment no later than 35 calendar days post-completion of RT.

2.4 Organ Function Requirements

2.4.1 Adequate Bone Marrow Function Defined as:

* Peripheral absolute neutrophil count (ANC) ≥ 1000/mm3.
* Platelet count ≥ 100,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).
* Hemoglobin > 8 g/dL (may be transfused).

2.4.2 Adequate Renal Function Defined as

* Creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73 m2 OR
* Maximum serum creatinine based on age/gender as follows: 10 to < 13 yrs=1.2 mg/dL for males and females. 13 to < 16 yrs=1.5 mg/dL for males and 1.4 mg/dL for females.

2.4.3 Adequate Liver Function Defined as:

* Total bilirubin must be ≤ 1.5 × institutional ULN.
* AST(SGOT)/ALT(SGPT) < 3 × institutional ULN.
* Alkaline Phosphatase < 3 × institutional ULN. 2.4.4 Informed consent: All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

1. Pregnancy or Breast-Feeding: Pregnant or breast-feeding women will not be entered on this study due to unknown potential risks of fetal and teratogenic adverse events as seen in animal studies. Pregnancy tests must be obtained in girls who are post-menarchal. Patients of childbearing or child fathering potential must agree to use one highly effective method of contraception while being treated on this study and for 3 months after completing therapy. A woman is considered of childbearing potential if she is fertile, following menarche and until becoming post-menopausal unless permanently sterile. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient. A man is considered fertile after puberty unless permanently sterile by bilateral orchidectomy. Male participants should refrain from sperm donation throughout the duration of treatment and for 3 months after completion of therapy.

   A highly effective contraception method is defined as one that results in a low failure rate (<1% per year) when used consistently and correctly. The following are considered highly effective contraception methods:
   * Combined estrogen and progesterone containing hormonal contraception associated with inhibition of ovulation.
   * Progesterone-only hormonal contraception associated with inhibition of ovulation.
   * Intra Uterine Device (IUD).
   * Intra uterine hormone releasing system.
   * Bilateral tubal occlusion.
   * Vasectomized partner.
   * Sexual abstinence (avoiding heterosexual intercourse).
   * The following contraceptive measures are NOT considered effective:

     * Progesterone-only hormonal contraception (birth control pill) that that does NOT stop ovulation.
     * Male or female condom with or without spermicide.
     * Cap, diaphragm, or sponge with spermicide.
2. Using the following types of concomitant medications:

   * Corticosteroids: Patients receiving corticosteroids are eligible. The use of corticosteroids must be reported.
   * Investigational Drugs: Patients who are currently receiving another investigational drug are not eligible.
   * Anti-cancer Agents: Concurrent anti-cancer agents are not allowed with the exception of temozolomide given concurrently with RT and as post RT maintenance therapy.
   * Anticonvulsants: Patients who are receiving enzyme inducing anticonvulsants that are strong inducers of CYP3A4/5 are not eligible.
   * Strong CYP3A4/5 inducers: Patients who are receiving strong inducers of CYP3A4/5 are not eligible. Strong inducers of CYP3A4/5 should be avoided from 14 days prior to or 5 half-lives (whichever is longer) enrollment to the end of the study.
   * Patients who are receiving medications known to prolong QTc interval are not eligible
   * Selective serotonin reuptake inhibitors (SSRIs) such as citalopram (Celexa), escitalopram (Lexapro), fluoxetine (Prozac), fluvoxamine (Luvox), paroxetine (Paxil), sertraline (Zoloft) should be used with caution but are not contraindicated.
   * Anticoagulants: patients who are receiving therapeutic anticoagulation with warfarin are not eligible.
3. Other Criteria

   * Infection: Patients who have an uncontrolled infection are not eligible.
   * Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study are not eligible.
   * Patients with known clinically significant active malabsorption syndrome or other condition that could affect absorption are not eligible.
   * Patients with malignancy related to HIV or solid organ transplant: known history of HIV, HBV surface antigen positivity or positive HCV antibody are not eligible. Viral testing is not required unless clinically indicated in patients without a known history.
   * Patients with prior or ongoing clinically significant illness, medical or psychiatric condition, that, in the investigator's opinion, could affect the safety of the subject, or could impair the assessment of study results are not eligible.
   * Patients with any prior solid organ transplant are not eligible.
   * Patients with secondary/radiation-related HGG are not eligible.
   * Patients with metastatic/disseminated HGG who have received CSI are not eligible.

Ages: 12 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2035-06 (Estimated)

PRIMARY OUTCOMES:
Establish the RP2D of Olutasidenib and Temozolomide (Feasibility cohort) | Completion of cycle 1 (28 days) for 6-24 patients
  To identify the dose of olutasidenib that is feasible when given post-RT in combination with temozolomide as maintenance therapy in pediatric and young adult patients newly diagnosed with IDH1-mutant high-grade glioma
Assess Progression-Free Survival (PFS) in Grade 3 IDH1-mutant Astrocytoma (Stratum A) | From date of diagnosis until date of Progressive Disease or death due to any cause or date of last follow-up, assessed up 24 months
  To assess the post-RT efficacy of olutasidenib in newly diagnosed patients with WHO Grade 3 IDH1-mutant Astrocytoma treated with maintenance olutasidenib and temozolomide for 13 cycles followed by 13 cycles of single agent olutasidenib compared to molecularly-stratified and matched historical controls
Maximum plasma concentration [Cmax] of Olutasidenib | From Day 1 of treatment until date of first documented progression or date of death from any cause, whichever comes first, assessed up to 24 months
  To characterize the plasma pharmacokinetic (PK) properties of olutasidenib in pediatric patients (e.g., 12 to < 18 years of age), administered in combination with temozolomide (first year) and as single agent (second year) as maintenance chemotherapy by measuring the Maximum Concentration [Cmax] and Area Under the Curve (AUC) of olutasidenib in plasma (All strata).

SECONDARY OUTCOMES:
Evaluate objective response rate (ORR) in HGG (All Strata) | From day 1 of protocol treatment through 30 days following end of protocol treatment
  Evaluate the radiographic objective response rate (ORR) defined as complete response (CR) + partial response (PR) in pediatric and young adult patients newly diagnosed with IDH1-mutant HGG treated with post-RT olutasidenib with temozolomide.
Evaluate Health-Related Quality of Life Outcomes (All Strata) | From pre-maintenance (2 weeks before the first cycle), and at the start of even numbered cycles (each cycle is 28 days) and at the End of Treatment visit (can have up to 26 cycles)
  Evaluate health-related quality of life outcomes of pediatric and young adult patients newly-diagnosed with IDH1-mutant HGG treated with post-RT olutasidenib by patient and/or parent reporting at key timepoints in therapy using the patient reported outcomes measurement information system (PROMIS) survey.
  These survey systems report scores on a scale of 1(minimum) to 5 (maximum). The scores may reflect frequencies from "1-Never" to "5-Always" or levels of autonomy from "1-With no trouble" to "5-Not able to do". Scores are interpreted differently for the different outcome measures
Evaluate Overall Survival in IDH1-mutant Grade 3 Astrocytoma (Stratum A) | From date of diagnosis until date of death due to any cause or date of last follow-up, assessed up to 60 months
  Determine distribution of OS in pediatric and young adult patients newly-diagnosed with IDH1-mutant Grade 3 Astrocytoma treated with post-RT olutasidenib and temozolomide for 13 cycles followed by 13 cycles of single agent olutasidenib compared to molecularly-stratified and matched historical controls.(Stratum A)
Assess Progression-Free Survival in IDH1-mutant Grade 4 Astrocytoma (Stratum B) | From date of diagnosis until date of Progressive Disease or death due to any cause or date of last follow-up, assessed up 24 months
  To assess the post-RT efficacy of olutasidenib in newly diagnosed patients with WHO Grade 4 IDH1-mutant Astrocytoma treated with maintenance olutasidenib and temozolomide for 13 cycles followed by 13 cycles of single agent olutasidenib compared to molecularly-stratified and matched historical controls

CONTACTS AND LOCATIONS:
Overall Officials: Santosh Valvi, FRACP, MSc, Study Chair — Perth Children's Hospital; Nicholas G Gottardo, MB FRACP PhD, Study Chair — Perth Children's Hospital; Michael J Fisher, MD, Study Chair — Children's Hospital of Philadelphia; Maryam Fouladi, MD, Study Chair — Nationwide Children's Hospital
Locations (18):
- United States (10):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Susan Chi, Boston, Massachusetts
  - Duke University Health System, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Australia (3):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Perth Children's Hospital, Perth, Western Australia
- Canada (2):
  - The Hospital for Sick Children (SickKids), Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
- Hopp Children's Cancer Center at NCT Heidelberg (KiTZ), Heidelberg, Baden-Wurttemberg, Germany
- Princess Máxima Center, Utrecht, Netherlands
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No